CLINICAL TRIAL: NCT02596854
Title: Comparative Study of Conventional 1.5 and 3.0T MR Images With Synthetically Reconstructed MR Images
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 114-2015-GES-0056
Record Dates: First submitted 2015-10-21; First posted 2015-11-04 (Estimated); Results first posted 2017-11-06 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Clinical Indication for Brain MRI

STUDY DESIGN:
Intervention Model Description: A single group will be enrolled from the general imaging population using the scanner available at the investigational site (either 1.5T or 3.0T, based on site determination and not specified per protocol). All participants are assigned to a single group.
Masking Description: None used for this single group study.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neurological MRI (Experimental): Images acquired for post processing with synthetic software. This is a crossover design where all subjects receive the same imaging scan, and comparison is done between the raw conventional scan and post-processed images using the research software.
  Interventions: Device: Neurological MRI

INTERVENTIONS:
Device: Neurological MRI — Neurological MRI image collection

SUMMARY:
This study is being conducted for regulatory submission of the GE Healthcare MAGnetic resonance Image Compilation (MAGiC), a point-of-care synthetic MR reconstruction software for GE 1.5T and 3.0T MR scanners.

DETAILED DESCRIPTION:
This study is a prospective, blinded, multi-center multi-reader (MCMR) clinical trial that is statistically powered for non-inferiority of diagnostic image quality of synthetic MR versus conventional MR and collection of supporting radiologic findings and morphology data from radiologists that reflect anticipated clinical usage of synthetic MR technology.

The study consists of three parts:

1. Clinical MR acquisition,
2. synthetic MR post-processing at a GE facility, and
3. blinded image evaluation (BIE) of conventional and synthetic images for each subject.

The study will enroll eligible adult subjects with clinical indications for brain MRI that meet applicable site MR safety criteria and are not pregnant. The study consists of one visit, the subject's MRI scan, without additional follow-up. Results are expected to be representative of expected clinical usage of synthetic MAGiC MR technology in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

1. Be an adult 18 years of age or older;
2. Have clinical indication for MRI of the brain according to the site standard of care;
3. If female of childbearing potential (not surgically sterile or post-menopausal), be determined non-pregnant by a medically qualified investigator or demonstrated non-pregnant by negative urine pregnancy test;
4. Be able to hear and understand instructions without assistive devices;
5. Have necessary mental capacity to understand instructions be able to comply with protocol requirements;
6. Are able and willing to provide written informed consent by signing the informed consent form (ICF).

Exclusion Criteria:

Subjects will be excluded that:

1. Were previously enrolled in this evaluation;
2. Have metallic/conductive or electrically/magnetically active implants or attached medical devices (except for dental devices/fillings, surgical clips, and surgical staples) that could be unsafe for MRI;
3. Have contraindication(s) to MRI scanning per the routine MR Safety Screening policy of the investigational site;
4. Have severe trauma or pre-existing pathology that is expected to interfere with normal conduct of MR scanning or complete scanning of the brain;
5. Have medical condition(s) such as those requiring urgent medical care that, in the opinion of a physician Investigator, would prevent safe participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Maryland Medical Center, Baltimore, Maryland
  - Advanced Radiology Services, PC/Spectrum Health, Grand Rapids, Michigan
  - The Mount Sinai Hospital, New York, New York
  - Cornell University, New York, New York
  - Manhattan Diagnostic Radiology (RadNet), New York, New York
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A single arm of subjects was enrolled and analyzed. Scanner selection (1.5T or 3.0T) was based on availability at the site and assigned by the site. Only one arm assignment (neurological MRI population) was per-protocol.
Groups:
- Neurological MRI: Image acquired for post processing with synthetic software
  Neurological MRI: Neurological MRI image collection
Period: Overall Study
Arm/Group | Neurological MRI
Started | 117
Completed | 109
Not Completed | 8
Not completed — Withdrawn | 8

BASELINE CHARACTERISTICS:
Population: The baseline is for all 117 participants, regardless of completion/withdrawal status. Patients were consented to allow information collected up until the time of withdrawal to remain on study to protect the integrity of the trial data.
Arm/Group | Neurological MRI
Number analyzed (Participants) | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 107
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 53.1 [19 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 50
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 117
Static Field Strength of MRI Scans [Count of Participants; unit: Participants]
  1.5T Scans | 58
  3.0T Scans | 59

OUTCOME MEASURES:

1. Primary Outcome: Mean Diagnostic Image Quality Difference Between Conventional Versus Synthetic MR Utilizing a 5 Point Likert Scale
Description: Images were read by board-certified radiologists who reviewed each image and assessed it on a 5 Point scale (1=unacceptable, 2=poor image quality, 3=Acceptable, 4=Good, 5=Excellent) based on the quality of the image (eg, signal-to-noise, clarity of anatomic boundaries, and other parameters). The outcome was reported as the mean diagnostic image quality score difference (synthetic - conventional).
Time Frame: 1 day
Population: Clinical indication for MRI of the brain based on site standard of care. This is a crossover study design where all subjects are enrolled into a single group producing two data types. The hypothesis test is a function of conventional and post-processed image quality within this patient group (one value summarized for this single population).
Measure: Mean (Standard Deviation); unit: units on a 5-point scale
Arm/Group | Neurological MRI
Number analyzed (Participants) | 109
units on a 5-point scale | -0.335 (0.3522)
Statistical Analysis 1: Comparison: Neurological MRI; Non-inferiority of synthetic MR versus conventional commercial MR the hypothesis can be stated as H0: S ≤ -Δ and HA: S > -Δ; Test type: Non-Inferiority — α=0.025 with a margin of Δ=0.5 were used for non-inferiority testing; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustments were made for multiple comparisons; Median Difference (Net) = -0.428, 95% CI 2-sided [-0.428 to -0.269], Standard Error of Mean 0.3522 — Notably, no separate comparative statistical analysis was performed for the 1.5T and 3.0T subgroups, which were pooled for analysis. All patients underwent both synthetic MR and commercial conventional MR in a single arm; To mitigate possible bias, the hypothesis test was executed via pre-programmed SAS module, which does not show the data for individual synthetic and conventional group values. The data for these individual groups is thus not currently available as part of the study report held by the sponsor or submitted to FDA. Thus, this data cannot be presented without additional analysis (re-programming) of the original SAS used to perform the study. Data were only reported as the difference between synthetic - conventional to determine non-inferiority, and data for individual crossovers (synthetic vs. conventional) were not calculated.The raw conventional scan images and those post-processed with the research software were combined as pre-specified in the study protocol

ADVERSE EVENTS:
Arm/Group | Neurological MRI
All-Cause Mortality (participants affected / at risk) | 0/117
Serious Adverse Events (participants affected / at risk) | 0/117
Other Adverse Events (participants affected / at risk) | 2/117
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neurological MRI (N=117)
Moderate Claustrophobia (General disorders) | 1 (1)
mild anxiety (General disorders) | 1 (1) — anxiety

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No